CLINICAL TRIAL: NCT06774040
Title: A Phase IIa Open Label, Dose-Finding, Clinical Trial to Evaluate Safety, Tolerability and Preliminary Efficacy of Etrinabdione in Patients With Peripheral Arterial Disease (PAD)
Brief Title: Evaluation of Safety, Tolerability and Preliminary Efficacy of Etrinabdione in Patients With Peripheral Arterial Disease
Acronym: CLAUDIA
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VivaCell Biotechnology España (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Etrinabdione-PAD02
Record Dates: First submitted 2024-12-20; First posted 2025-01-14 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Arterial Disease
Keywords: Claudication; Arterial Occlusive Disease; Peripheral Artery Disease; Vascular Disease; Peripheral Vascular Disease; Chronic Limb Threatening Ischemia; Critical Limb Ischemia
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Arterial Occlusive Diseases; Vascular Diseases; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia | interventions — BID protein, human

STUDY DESIGN:
Intervention Model Description: The trial will start with the lower dose (25 mg BID). When the 12 patients have been treated for 3 months and the PK and safety data are evaluated by the regulatory authority, the Sponsor and the site investigators, the high dose (50 mg BID) will be released.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low dose (Experimental): 25 mg BID
  Interventions: Drug: Etribnabdione 25 mg BID
- High dose (Experimental): 50 mg BID
  Interventions: Drug: Etribnabdione 50 mg BID

INTERVENTIONS:
Drug: Etribnabdione 25 mg BID — The trial will start with the lower dose. When the 12 patients have been treated for 3 months and the PK and safety data are evaluated by the regulatory authority, the Sponsor and the site investigators, the high dose (50 mg BID) will be released.
  Arms: Low dose
Drug: Etribnabdione 50 mg BID — The treatment will start when the regulatory authority, the sponsor and the site investigators have reviewed the low dose safety and pharmacokinetics data.
  Arms: High dose

SUMMARY:
The goal of this clinical trial is to study the safety and tolerability of Etrinabdione in adult patients with peripheral arterial disease. It will also learn about the preliminary efficacy of Etrinabdione. The main questions it aims to answer are:

Has Etrinabdione an acceptable safety/tolerability profile during 12 months?

Do the patients show any improvement in any of the tests included in the protocol for this disease?

Researchers will test first the low dose of Etrinadione. If the product is safe at 3 months, the high dose can start.

Participants will:

Take Etrinabdione twice a day for 12 months. Visit the clinic once every 4 weeks for checkups and tests.

DETAILED DESCRIPTION:
This is a single center, open-label Phase IIa clinical study. The study will be conducted with 2 treatment arms 25 mg BID and 50 mg BID.

The study consists of a Screening Period, a Treatment Period, and a Follow-up Period. Total duration 14 months.

Subjects who meet the inclusion criteria and do not meet the exclusion criteria at screening will start with the lower dose (25 mg BID). When the 12 patients have been treated for 3 months and the PK and safety data are evaluated by the regulatory authority, the Sponsor and the site investigators, the high dose (50 mg BID) will be released.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent and capable of understanding and complying with the protocol;
* Subjects classified as critical limb ischemia (CLI) Rutherford Category 2 or 3 (moderate or severe) claudication;
* Diabetes mellitus type 2 with HbA1c < 9%;
* In case of treatment for PAD, the subject is controlled on medical therapy indicated for CLI;
* A female patient is eligible to participate if she is not pregnant, not breastfeeding, and agrees to use a highly effective method of contraception;
* A male patient with a female partner of childbearing potential is eligible if he agrees to use acceptable method of contraception.

Exclusion Criteria:

* Planned surgical or endovascular revascularization on the index leg within the next 12 months;
* Failed surgical or endovascular revascularization on the index leg within 10 days prior to screening;
* Amputation at or above the talus on the index leg;
* Planned major amputation within the first month after screening;
* On the index leg, use of concomitant wound treatments not currently approved for ischemic wound-healing within 30 days prior to screening or plans to initiate new treatments to the index leg during the trial;
* Uncontrolled or untreated proliferative retinopathy;
* Blood clotting disorder not caused by medication;
* Severe hypertension according to the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure;
* Evidence of moderate to severe hepatocellular dysfunction;
* Positive test for human immunodeficiency virus 1 (HIV 1), HIV 2, hepatitis B virus (HBV), hepatitis C virus (HCV) or Treponema Pallidum;
* Subjects who may not be healthy enough to successfully complete all protocol requirements, or who are not expected to survive more than 12 months, or in whom results may be particularly difficult to assess.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Treatment Emergent Adverse Events (TEAEs) | 13 months
  This safety outcome combines the measure of the number of subjects experiencing adverse events (AEs), the nature and severity of those AEs and their relationship to the study treatments.

SECONDARY OUTCOMES:
Vascularization | Baseline, 6 and 12 months
  The angiogenesis induced by Etrinabdione treatment will be assessed by the evaluation of the peripheral arterial system of affected limbs by computed tomography angiography.
Absolute claudication time | Baseline, 3, 6 and 12 months
  The claudication time will be quantitatively measured by standardized treadmill test using a graded exercise protocol.
Hemodynamic | Baseline, 3, 6 and 12 months
  The Ankle/Brachial Index (ABI) is a diagnostic measure used to assess blood flow and detect potential vascular abnormalities. It will be calculated as the ratio of systolic blood pressure at the ankle level (posterior tibial artery or pedia) divided by the systolic blood pressure obtained on the arm (humeral artery).
Stenosis | Baseline, 3, 6 and 12 months
  Doppler ultrasound will be performed in the affected lower limbs at the level of the common femoral artery, superficial femoral artery, popliteal artery, posterior tibial artery and pedia artery.
Disease specific quality of life questionnaire (VascuQoL-6) | Baseline, 3, 6 and 12 months
  The questionnaire includes 6 questions with 4 possible answers, scoring from 1 to 4. The lower the score, the worse the patient's perceived quality of life.
Tissue oxigenation | Baseline, 3, 6 and 12 months
  Measure the local oxygen released from the capillaries through the skin by transcutaneous oximetry.

OTHER OUTCOMES:
Pharmacokinetic profile of Etrinabdione in terms of maximum observed plasma concentration (Cmax). | pre-dose and 3 hours post dose) at Day 1 and months 1, 3, 6, 12, and 13 months.
  The point of maximum concentration of Etrinabdione in plasma.
Pharmacokinetic profile of Etrinabdione in terms of time to peak drug concentration (Tmax). | pre-dose and 3 hours post dose) at Day 1 and months 1, 3, 6, 12, and 13 months.
  The time of Etrinabdine to reach its maximum concentration in the body after administration
Pharmacokinetic profile of Etrinabdione in terms of area under the plasma concentration-time curve (AUC). | pre-dose and 3 hours post dose) at Day 1 and months 1, 3, 6, 12, and 13 months.
  Total systemic exposure to Etrinabdione.
Determination of potential accumulation of Etrinabdione. | pre-dose and 3 hours post dose) at Day 1 and months 1, 3, 6, 12, and 13 months.
  Etrinabdione plasma through level.
Change in blood levels of disease/mechanism of action biomarkers measured by proximity extension assay and next-generation sequencing. All levels of plasma proteins will be provided in normalized protein expression units (NPX). | Day 1 and months 1, 3, 6, 12, and 13 months.
  von Willebrand factor, Angiogenin, EPO, HGF, VEGF, FGF-2, PDGF, Endoglin, Endothelin-1, IL-1, TNFa, IL-6, IL-17, ICAM-1, IL-18, Proteinase-activated receptor 1, Angiopoietin-1, Endothelial cell-specific molecule 1, IL-18 and MCP1

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Reina Sofía, Córdoba, Spain

REFERENCES:
- [Background] Garcia-Martin A, Prados ME, Lastres-Cubillo I, Ponce-Diaz FJ, Cerero L, Garrido-Rodriguez M, Navarrete C, Pineda R, Rodriguez AB, Munoz I, Moya J, Medeot A, Moreno JA, Chacon A, Garcia-Revillo J, Munoz E. Etrinabdione (VCE-004.8), a B55alpha activator, promotes angiogenesis and arteriogenesis in critical limb ischemia. J Transl Med. 2024 Nov 6;22(1):1003. doi: 10.1186/s12967-024-05748-w. PMID 39506809
- See also: Company website — https://vivacellspain.com/